CLINICAL TRIAL: NCT00043953
Title: A Phase II Study of Lopinavir/Ritonavir in Combination With Saquinavir Mesylate or Lamivudine/Zidovudine to Explore Metabolic Toxicities in Antiretroviral HIV-Infected Subjects
Brief Title: Lopinavir/Ritonavir in Combination With Saquinavir Mesylate or Lamivudine/Zidovudine to Explore Metabolic Toxicities in Antiretroviral HIV-Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M01-384
Record Dates: First submitted 2002-08-15; First posted 2002-08-19 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections
Keywords: treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Saquinavir; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Saquinavir mesylate
Drug: Lamivudine/zidovudine

SUMMARY:
The objectives of this study are to explore the metabolic toxicities associated with lopinavir/ritonavir (LPV/r) plus saquinavir mesylate (INV) versus LPV/r plus Combivir in antiretroviral naïve subjects and to assess the overall safety, tolerability and efficacy of LPV/r plus INV versus LPV/r plus Combivir in antiretroviral naïve subjects and to assess the pharmacokinetics of 400 mg INV taken twice a day (BID), 600 mg INV BID and 800 mg INV BID in combination with 400 mg lopinavir/100 mg ritonavir plus 150 mg lamivudine/300 mg zidovudine BID.

ELIGIBILITY:
Inclusion Criteria:

* Subject is naïve to antiretroviral treatment (subjects may not have more than 7 days of any antiretroviral treatment).
* Subject is at least 18 years of age, inclusive.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:condoms, sponge, foams, jellies, diaphragm or intrauterine device(IUD), a vasectomized partner, total abstinence from sexual intercourse
* If female, the results of a urine pregnancy test performed at screening (urine specimen obtained no earlier than 28 days prior to study drug administration) is negative.
* Subject is not breast-feeding.
* Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness.
* Subject has no significant history of cardiac, renal, neurologic, psychiatric, oncologic, endocrinologic, metabolic or hepatic disease that would in the opinion of the investigator adversely affect his/her participating in this study.
* Subject does not require and agrees not to take any of the following medications for the duration of the study: midazolam, triazolam, terfenadine, astemizole, cisapride, pimozide, propafenone, flecainide, certain ergot derivatives (ergotamine, dihydroergotamine, ergonovine, and methylergonovine), rifampin, lovastatin, simvastatin, and St. John's wort.
* Subject agrees not to take any medication during the study, including over-the-counter medicine, alcohol or recreational drugs without the knowledge and permission of the principal investigator.
* Subject has not been treated for an active AIDS-defining opportunistic infection within 30 days of screening.
* Subject has a plasma HIV RNA level of greater than 400 copies/mL at screening.
* Subject agrees to take all doses of the study drug from the bottles provided by the sponsor (rather than other containers, i.e., "pill box").
* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.

Exclusion Criteria:

* Subject has a history of an allergic reaction or significant sensitivity to LPV/r, INV or Combivir.
* Subject has a history of substance abuse or psychiatric illness that could preclude adherence with the protocol.
* Screening laboratory analyses show any of the following abnormal laboratory results:

  * Hemoglobin ≤ 10.0 g/dL
  * Absolute neutrophil count ≤ 1000 cells/µL
  * Platelet count ≤ 50,000 per mL
  * ALT or AST ≥ 3.0 x Upper Limit of Normal (ULN)
  * Creatinine ≥ 1.5 x Upper Limit of Normal (ULN)
* Subject has received any investigational drug within 30 days prior to study drug administration.
* For any reason, subject is considered by the investigator to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-08

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV RNA level below 50 copies/mL | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A da Silva, M.D., Study Director — Associate Medical Director, Antiviral Global Project Team
Locations (11):
- United States (9):
  - AHF Research, Los Angeles, California
  - Pacific Horizon Medical Group, San Francisco, California
  - Stephen Becker, MD, San Francisco, California
  - Harbor UCLA, Research & Education Institute, Torrance, California
  - Community Research Initiative of New England, Boston, Massachusetts
  - Community Research Initiative of New England, Springfield, Massachusetts
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
- Canada (2):
  - University of Ottawa at the Ottawa Health Research Institute, Ottawa
  - University of Ottawa Health Research Institute, Ottawa